CLINICAL TRIAL: NCT00107588
Title: Contingency Management for Marijuana Dependence
Brief Title: Marijuana Treatment Project - 3
Acronym: MTP-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-12728-06; R01DA012728-06 (NIH); R01-12728-06
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Marijuana Dependence
Keywords: marijuana dependence; self-efficacy; coping skills; attendance; marijuana abstinence
MeSH Terms: conditions — Marijuana Abuse | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reinforcement for homework completion (Experimental)
  Interventions: Behavioral: Reinforcement for homework completion
- Reinforcement for Abstinence (Active Comparator)
  Interventions: Behavioral: Reinforcement for Abstinence
- Case Management (Active Comparator)
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Reinforcement for homework completion — Provides contingent reinforcement for engaging in homework activities designed to enhance coping skills
  Arms: Reinforcement for homework completion
Behavioral: Reinforcement for Abstinence — Provides contingent reinforcement for submitting marijuana-free urine specimen
  Arms: Reinforcement for Abstinence
Behavioral: Case Management — Will control for the effect of therapist-client contact by providing supportive case management as an active control condition.
  Arms: Case Management

SUMMARY:
The goal of this research is to improve treatment outcome for marijuana-dependent individuals. The current study builds on the findings of our prior NIDA-funded marijuana treatment study in which improved client outcomes were associated with greater treatment attendance, greater client self-efficacy, and greater use of coping skills. We will use a contingency management paradigm to provide tangible reinforcement for completing homework assignments that are designed to enhance coping skills. It is anticipated that this will result in greater homework compliance, leading to greater self-efficacy regarding one's ability to cope with high-risk situations. Improved self-efficacy will enhance the likelihood of employing coping skills in high-risk situations, thereby increasing the probability of achieving and maintaining abstinence.

DETAILED DESCRIPTION:
Participants will receive an intervention combining one session of motivational enhancement therapy with eight sessions of cognitive-behavioral coping skills therapy (MET+CBT). A contingency management procedure will be added to this intervention, providing reinforcement for completion of homework, as verified by call-ins to an Interactive Voice Recording (IVR) system. Outcomes will be compared to an MET+CBT intervention in which reinforcement will be provided for marijuana-free urine specimens, and to a control group that receives Case Management. Recruitment of 234 marijuana-dependent participants will occur over a three-year period. They will be randomly assigned to one of the three 9-session interventions. Treatment will be individual, manualized, and provided on an outpatient basis. Pretreatment assessments will obtain baseline data; follow-up assessments at three-month intervals for one year will evaluate marijuana use outcomes, other drug or alcohol use, and psychosocial functioning. It is anticipated that the intervention in which completion of homework is reinforced will result in the best outcomes. The mechanisms by which the interventions result in behavior change will be the specific focus of attention in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis dependence
* Willing to accept random assignment to interventions

Exclusion Criteria:

* Current dependence on alcohol or other drugs
* Problems that require inpatient hospitalization
* Reading ability below fifth grade level
* Lack of reliable transportation to treatment
* Excessive commuting distance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-02; Primary Completion 2011-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Marijuana abstinence | One-year follow-up period
Self-efficacy, use of coping skills, and treatment attendance | During 2-month treatment period

SECONDARY OUTCOMES:
Continuous abstinence will be predicted by (a) treatment attendance; (b) posttreatment self-efficacy for coping; and (c) use of coping skills | One-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States